CLINICAL TRIAL: NCT03228511
Title: Evaluation of Endoscopic-assisted Microsurgical Removal of Cerebellopontine Angle Lesions
Brief Title: Endoscopic-assisted Microsurgical Removal of Cerebellopontine Angle Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammad Tamam, Principal invistigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Easpost fossa
Record Dates: First submitted 2017-07-18; First posted 2017-07-25 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Cerebellopontine Angle Tumor
MeSH Terms: conditions — Neuroma, Acoustic | interventions — Endoscopes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Formerly Arm Label (Experimental)
  Interventions: Device: endoscope

INTERVENTIONS:
Device: endoscope — It is a Prospective descriptive hospital based clinical study to determine the value of introduction of endoscope after microscopic excision of cerebello-pontine angle lesions

SUMMARY:
It is a Prospective descriptive hospital based clinical study to determine the value of introduction of endoscope after microscopic excision of cerebello-pontine angle lesions to estimate the following :

1. Intraoperative judgement of lesions excision, residual parts, visualization and operative corridor pre and after endoscope introduction.
2. Post-operative tumor control confirmed comparison between pre and postoperative MRI.
3. Postoperative complications, advantages and disadvantages compared with these when use pure microscopic excision from the literature

ELIGIBILITY:
Inclusion Criteria: cerebellopontine angle lesions

* meningeoma.
* vestibular schwannoma.
* arachnoid cyst.
* petroclival meningeoma.

Exclusion Criteria:

* trigeminal neuralgia.
* facial neuralgia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
post operative residual tumor | 1 week
  post operative MRI will be done and will be compared with the preoperative one to determine if complete excision was done or if there is residual parts